CLINICAL TRIAL: NCT06049446
Title: Combining Contrast-Enhanced Mammography and Radio-active Free Magnetic Seed Localization of Non-palpable Breast Tumors: A Feasibility Study
Brief Title: Combining CEM and Magnetic Seed Localization of Non-Palpable Breast Tumors
Acronym: CEMMAG
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: CEMMAG
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: Breast neoplasms; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients receiving seed localization: Patients receiving seed localization
  Interventions: Device: Pintuition

INTERVENTIONS:
Device: Pintuition — Magnetic seed localization

SUMMARY:
Rationale: Breast cancer patients are increasingly treated with neoadjuvant chemotherapy for various reasons. These women receive chemotherapy before any surgery is performed. Many of these tumors need preoperative seed localization to help guide the surgeons to the site of the tumor within the breast. The interest is shifting towards to use of non-radioactive seeds, such as the magnetic seeds used in this study. A drawback of these seeds is the fact that they cause large susceptibility artifacts on (magnetic!) MRI of the breast. Breast MRI is the most accurate modality to monitor response to therapy of these women. CEM, an emerging breast imaging technique, has shown to achieve comparable results with regard to response monitoring but uses no magnetic fields. Hence, CEM might be an attractive alternative response monitoring tool in patients treated with neoadjuvant chemotherapy and having a magnetic seed a surgical marker. To this point, however, no study in humans has confirmed that this is indeed the case.

Objective: To test whether the use of magnetic localization seeds causes image artifacts on CEM.

Study design: Observational feasibility study.

Study population: Women (>18 years) able to provide written informed consent and recently diagnosed with (non-palpable) breast cancer or ductal carcinoma in situ (DCIS), who are primarily treated with surgery.

Intervention (if applicable): Image-guided placement of a magnetic seed (Sirius Pintuition) prior to surgery, including control imaging to confirm the correct location of the seed relative to the breast abnormality. In usual patient care this is performed with full-field digital mammography (FFDM), but in this study this control image will be performed with the system in 'contrast-enhanced mammography' or CEM mode, but without using intravenous administration of iodinated contrast agent because the purpose is not repetition of diagnostic imaging, but to rule out any artifacts caused by the seed on CEM. The investigators estimate to include twenty patients to confidently test the hypothesis that magnetic seeds do not cause disturbing artifacts on CEM examinations.

Main study parameters/endpoints: The primary study aim will be to test whether the magnetic seeds caused any disturbing artifacts on CEM images. As secondary study, the investigators will document technical success rate of seed deployment and retrieval during surgery, including the assessment of the surgical margins (positive or negative).

DETAILED DESCRIPTION:
Rationale: Breast cancer patients are increasingly treated with neoadjuvant chemotherapy for various reasons. These women receive chemotherapy before any surgery is performed. Many of these tumors need preoperative seed localization to help guide the surgeons to the site of the tumor within the breast. In many hospitals, a radioactive I-125 seed is used for this purpose, which has several disadvantages, such as a slight increase in radiation dose and extensive administrative regulations to monitor the location of the seed at any time (required by law). This administrative work is time consuming, elaborate and prone to errors. Therefore, interest is shifting towards to use of non-radioactive seeds, such as the magnetic seeds used in this study. A drawback of these seeds is the fact that they cause large susceptibility artifacts on (magnetic!) MRI of the breast. Breast MRI is the most accurate modality to monitor response to therapy of these women. CEM, an emerging breast imaging technique, has shown to achieve comparable results with regard to response monitoring but uses no magnetic fields. Hence, CEM might be an attractive alternative response monitoring tool in patients treated with neoadjuvant chemotherapy and having a magnetic seed a surgical marker. To this point, however, no study in humans has confirmed that this is indeed the case.

Objective: To test whether the use of magnetic localization seeds causes image artifacts on CEM.

Study design: Observational feasibility study. Study population: Women (>18 years) able to provide written informed consent and recently diagnosed with (non-palpable) breast cancer or ductal carcinoma in situ (DCIS), who are primarily treated with surgery.

Intervention (if applicable): Image-guided placement of a magnetic seed (Sirius Pintuition) prior to surgery, including control imaging to confirm the correct location of the seed relative to the breast abnormality. In usual patient care this is performed with full-field digital mammography (FFDM), but in this study this control image will be performed with the system in 'contrast-enhanced mammography' or CEM mode, but without using intravenous administration of iodinated contrast agent because the purpose is not repetition of diagnostic imaging, but to rule out any artifacts caused by the seed on CEM. The investigators estimate to include twenty patients to confidently test the hypothesis that magnetic seeds do not cause disturbing artifacts on CEM examinations.

Main study parameters/endpoints: The primary study aim will be to test whether the magnetic seeds caused any disturbing artifacts on CEM images. For this purpose, two radiologists will score the images for the presence of any artifacts and if present, if these are to such an extent that they would hamper diagnostic evaluation of the images. The radiologists will assess the images independently first, and consensus opinion is formed should any discrepancies occur in their judgement. As secondary study, the investigators will document technical success rate of seed deployment and retrieval during surgery, including the assessment of the surgical margins (positive or negative).

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: The burden and risk for participating subjects are very small. In regular care, a radioactive I-125 seed is placed in the breasts of these women, checking the position with (conventional) FFDM. For this purpose, the iodine seed is replaced with a (radioactive-free) magnetic seed (Sirius Pintuition). The latter did not show any relevant imaging artifacts prior to this study in imaging phantoms (i.e., chicken breasts containing magnetic seeds). Therefore, the investigators feel confident that these seeds will not show artifacts on clinical CEM image, but this needs to be confirmed before additional studies regarding the clinical application of CEM and magnetic seeds combined can be safely performed. The only additional disadvantage for participants is the slight increased radiation dose of the (extra) high-energy image CEM image, which is an increased radiation dose to the breasts of 50-80%. However, these women are all diagnosed with breast cancer requiring adjuvant radiotherapy, which uses radiation doses much, much higher than a single mammographic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Included are non-pregnant women (>18 years of age),
* Recently diagnosed with non-palpable invasive breast cancer or DCIS, requiring primary surgical treatment.
* Only women able to provide written informed consent will be considered for this study.

Exclusion Criteria:

- Excluded are women not meeting the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with breast cancer
Study Population: For this purpose, women meeting the inclusion criteria (see paragraph 4.2) will be asked to participate in this study. If they consent, the regular localization using a I-125 marker will be replaced by the magnetic seed, but the remainder of the procedure of implantation is identical (image guided placement using local anesthesia). Normally, a conventional (full-field digital) mammogram is acquired to establish the (correct) position of the marker with respect to the lesion of interest. For this study, we will select the 'CEM' mode instead of 'FFDM' mode on the mammography unit. This will result in having a standard CEM examination. Since the images are intended to check for artifacts caused by the seed, we decided not to administrate iodinated contrast agent to reduce patient's burden (as this would require catheter placement and contrast administration, potentially resulting in complications such as infection, hematoma, and hypersensitivity reactions to the contrast used). A low-ener
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Assessment of image artifacts | 1 day
  Main study endpoint will be the assessment of the occurrence of image artifacts, which will be scored by blinded radiologists in the following way: if there are any artifacts present in the image (yes/no) and caused by the magnetic seed
Influence of image artifacts | 1 day
  If primary outcome measure #1 is answered with yes: are the artifacts influencing the overall image quality (yes/no)?

SECONDARY OUTCOMES:
Technical success rate of seed deployment | 1 month
  The investigators will evaluate how often the seed deployment was considered succesful (in %)
Technical success rate of see retrieval during surgery | 1 month
  The investigators aim to evaluate how often the seed could not be retrieved during surgery of the breast (in %)
Surgical outcome | 1 month
  The investigators aim to study how often the surgical margins were not radical, i.e. still contained invasive breast cancer or DCIS (in %)

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD is not expected for this study nor its outcomes.